CLINICAL TRIAL: NCT05504902
Title: Vibrotactile Coordinated Reset for the Treatment of Advanced Parkinson's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vivek P. Buch, Protocol Director, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 66691
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Non-invasive
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Vibrotactile Coordinated Reset (vCR) (Experimental): Vibrotactile Coordinated Reset delivers vibratory stimulation to the fingertips of each hand. A specific pattern of vibration to each fingertip is delivered which theoretically disrupts abnormal synchrony in the brain.
  Interventions: Device: Vibrotactile coordinated reset

INTERVENTIONS:
Device: Vibrotactile coordinated reset — The purpose of this study is to test the efficacy of vibrotactile coordinated reset stimulation on human subject participants with Advanced stage Parkinson's disease

SUMMARY:
The purpose of our study is to evaluate Vibrotactile Coordinated Reset stimulation (vCR) and its effects on advanced stage Parkinson's symptoms. VCR will be administered with a device called the Stanford CR Glove. vCR is expected to provide patients with a non-invasive alternative to the most widely used treatments such as levodopa and or deep brain stimulation. Patients will be followed for two years.

DETAILED DESCRIPTION:
This study involves gentle vibrations delivered to the finger-tips which have been shown in pilot studies to be effective in reducing motor symptoms associated with Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of enrollment: 18 years of age or older
2. Idiopathic Parkinson's Symptoms between hoehn and yahr stages 2 to 4
3. Fluent in English
4. If patient is on medication that affects brain function or alters EEG activity, the patient must feel comfortable going off this medication prior to EEG recording
5. Appropriate social support if required during an off state.
6. Comfortable with technology; can use a computer, check email, and access the internet; can initiate and engage in a virtual meeting for training and monitoring purposes.
7. Feels comfortable going off PD related medication during in person study visits.
8. Lives in the United States

Exclusion Criteria:

1. Any significant neuro-psychiatric problems, including acute confusional state, ongoing psychosis, or suicidal tendencies
2. Any current drug or alcohol abuse.
3. Participation in another drug, device, or biologics trial concurrently or within the preceding 30 days. Any other trial participation should be approved by the Principal Investigators.
4. Pregnancy, breast-feeding or wanting to become pregnant
5. Physical limitations unrelated to PD that would affect motor ratings
6. Craniotomy
7. Brain surgery
8. Patient is unable to communicate properly with staff (i.e., severe speech problems)
9. Excessive drooling
10. A type of hair style that would impede the use of an EEG cap
11. Sensory abnormalities of the fingertips
12. Patient is taking a medication that may cause significant withdrawal effects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Movement Disorders Society Unified Parkinson's Disease Rating Scale Part 3 (MDS-UPDRS III) off medication | Baseline, 6 months, 12 months, 18 months, 24 months
  This scale measures motor ability within Parkinson's patients. For part 3, the scales minimum values is 0 and max value is 132. Higher scores indicate more impaired motor ability, while lower scores indicate less impaired motor ability. A score of 0 indicates no motor impairment. This assessment is performed while participants are off Parkinson's-related medication.

SECONDARY OUTCOMES:
Levodopa equivalent daily dose (LEDD) | Baseline, 24 months
  LEDD is calculated as a daily sum of levodopa in each Parkinson's medication
Parkinsons disease quality of life questionnaire-39 (PDQ-39) | Baseline, 6 months, 12 months, 18 months, 24 months
  The PD Quality of Life Questionnaire-39 (PDQ-39) is a self-report questionnaire that examines health related difficulties specific to PD in eight quality of life categories within the last month. Items are grouped into eight scales that are scored by expressing summed item scores as a percentage score ranging between 0 and 100, with higher % indicating more health problems.
Freezing of Gait Questionnaire (FOG) | Baseline, 6 months, 12 months, 18 months, 24 months
  The Freezing of Gait questionnaire (FOG) assesses severity unrelated to falls in patients with Parkinson's Disease (PD), FOG frequency, disturbances in gait, and relationship to clinical features conceptually associated with gait and motor aspects (e.g., turning). The FOG is comprised of 6 questions measured on a 0 to 4 scale (where 0 is normal and 4 represents severe abnormalities). The scores are summed together with 0 representing the best possible score and 24 representing the worst possible score.
Movement disorders unified Parkinson's rating scale (MDS-UPDRS) part 1 | Baseline, 6 months, 12 months, 18 months, 24 months
  The MDS-UPDRS part 1 focuses on non-motor symptoms, such as dementia, depression, and psychosis. The total summed score ranges from 0-52 with higher scores indicating increased non-motor impairment.
Movement disorders unified Parkinson's rating scale (MDS-UPDRS) part 2 | Baseline, 6 months, 12 months, 18 months, 24 months
  The MDS-UPDRS part 2 focuses on the patient's ability to perform daily motor activities including dressing, grooming, and using utensils. The total summed score ranges from 0-52 with higher scores indicating increased daily motor impairment.
Movement disorders unified Parkinson's rating scale (MDS-UPDRS) part 4 | Baseline, 6 months, 12 months, 18 months, 24 months
  The MDS-UPDRS 4 focuses on Measures the complications of treatment, e.g. dyskinesias and motor fluctuations. The total summed score ranges from 0-24 with higher scores indicating increased motor complications.
Communicative Participation Item Bank (CPIB; Short Form) | Baseline, 6 months, 12 months, 18 months, 24 months
  The CPIB is a questionnaire that measures speech complications. The questionnaire is scored from 0 to 30, with a higher score indicating increased speech difficulties.
Voice Handicap Index (VHI-10) | Baseline, 6 months, 12 months, 18 months, 24 months
  This questionnaire can be filled out by patients and assesses the impact that voice problems and limitations have on the individual's overall daily function. Questionnaire is scored from 0 to 40, with a higher score indicating increased speech difficulties.
Spontaneous EEG beta band power | Baseline, 6 months, 12 months, 18 months, 24 months
  Patients will be recorded while receiving vibrotactile stimulation. The Beta Band (13-30Hz) power spectral density (PSD) will be of interest. The units of the power spectral density are micro-Volts-squared per Hz. Increases in Beta band PSD are associated with motor impairment in Parkinson's disease, while decreases in the beta band are associated with motor improvement.
Parkinson's disease cognitive functional rating scale (PD-CFRS) | Baseline, 6 months, 12 months, 18 months, 24 months
  The PD-CFRS capture subjective daily functional cognitive decline among patients with Parkinson's disease over the past 2 weeks. The scale ranges from 0 to 24, with higher scores indicative of cognitive decline.
Vibratory threshold | Baseline, 6 months, 12 months, 18 months, 24 months
  Participants will be assessed for their perceptive threshold of vibration, or the lowest vibration amplitude perceived. This is determined by adjusting the amplitude of the experimental device.
Movement Disorders Society Unified Parkinson's Disease Rating Scale Part 3 (MDS-UPDRS III) on medication | Baseline, 6 months, 12 months, 18 months, 24 months
  This scale measures motor ability within Parkinson's patients. For part 3, the scales minimum values is 0 and max value is 132. Higher scores indicate more impaired motor ability, while lower scores indicate less impaired motor ability. A score of 0 indicates no motor impairment. This assessment is performed while participants are on Parkinson's-related medication.

OTHER OUTCOMES:
Quantitative Digitography Repetitive Alternating Finger Task (QDG-RAFT) | Baseline, 1 week, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months
  The QDG-RAFT requires participants to place their index and middle finger on adjacent keys of a digitography device. They are instructed to press and release each key in an alternating pattern, as fast and regularly as possible for thirty seconds, starting and stopping only when an auditory cue is heard. This is an exploratory measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States